CLINICAL TRIAL: NCT01179061
Title: Investigating the Inotropic Potential of Apelin in Healthy Volunteers and Patients With Chronic Stable Heart Failure
Brief Title: Investigating the Inotropic Potential of Apelin
Acronym: INO-apelin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Edinburgh (Other)
Responsible Party: Dr Gareth Barnes, University of Edinburgh
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 10/S1101/18
Record Dates: First submitted 2010-08-09; First posted 2010-08-10 (Estimated); Last update posted 2024-05-09 (Actual); Status verified 2010-08

CONDITIONS: Heart Failure
Keywords: Apelin; Heart failure; Pulmonary artery pressure; Inotropic; Diuretic
MeSH Terms: conditions — Heart Failure | interventions — Apelin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Apelin infusion (Experimental): 6 hour infusion of apelin peptide into circulation
  Interventions: Drug: Apelin
- Placebo (Placebo Comparator): Infusion of saline into systemic circulation
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Apelin — Cardiac index will be assess in patients through the 6hr infusion, using thoracic cardiac bioimpedance. Prior to starting the infusion there will be a 30 minute run in period to achieve a stable cardiac index. Thereafter the infusion will be started, with cardiac index assess every five minutes during the first hour. For each subsequent hour participants will be free to mobilise for the thirty minute periods, with cardiac index and systemic haemodynmics assess for the following thirty minutes.
  Additionally during the first hour pulmonary artery pressure will be estimated from pulmonary artery pressures assessed with echocardiography. This will be assessed at baseline with four further measurements during the first hour of infusion.
  Participants will be asked to void prior to the study starting, thereafter all urine will be collected during the course of the study. Relevant biochemical/humoral factors will be assessed in the urine.
  Arms: Apelin infusion
Drug: Placebo — As per apelin arm, however we will use a saline placebo infusion. All other aspects will remain the same.
  Arms: Placebo

SUMMARY:
The apelin-APJ system is a recently discover hormone system that has several important actions in the cardiovascular system. Apelin causes the heart pump with more force and also causes blood vessels to relax. Studies to date show that people with reduced pumping function of the heart have lower levels of apelin in the bloodstream compared to people with normal heart function. We have previously given apelin to healthy volunteers and people with reduced pumping function and this increases the heart's contraction. However, this has only been assessed over a short time period, around fifteen minutes, and we now want to know if this effect is seen over a longer period.

ELIGIBILITY:
Inclusion Criteria:

Healthy volunteers:

>18yrs

Heart failure patients;

* New York Heart Failure class II-IV
* Ejection fractional <35% or fractional shortening <20% within previous 6months.

Exclusion Criteria:

All subjects,

* Females of child bearing age not on adequate contraception
* Lack of informed consent
* Age <18yrs
* Current involvement in any other research study
* Systolic BP >190 or <100
* Malignant arrhythmias
* Renal or hepatic failure
* Haemodynamically significant aortic stenosis
* Severe or significant co-morbidity
* Pacemakers

Healthy volunteers

* Any regular medication
* Previous history of any cardiovascular disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2010-08; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
cardiac output | 6 hours
  We will assess, using thoracic bioimpedance cardiography, the change in cardiac output in response to apelin infusion

SECONDARY OUTCOMES:
Urine volume | 6 hours
  All urine will be collected during the studya and we will assess volume and relevant biochemical/humoral factors
Pulmonary artery pressure | 1 hour
  Using echocardiography we will estimate the pulmaonary artery pressure from pulmonary velocity and assess any change during the first hour of study.

CONTACTS AND LOCATIONS:
Locations (3):
- United Kingdom (3):
  - Clincial Research Facility, Royal Infirmary of Edinburgh, 51 Little France Cresc, Edinburgh
  - Gareth Barnes, Edinburgh
  - University of Edinburgh, Edinburgh

REFERENCES:
- [Derived] Barnes GD, Alam S, Carter G, Pedersen CM, Lee KM, Hubbard TJ, Veitch S, Jeong H, White A, Cruden NL, Huson L, Japp AG, Newby DE. Sustained cardiovascular actions of APJ agonism during renin-angiotensin system activation and in patients with heart failure. Circ Heart Fail. 2013 May;6(3):482-91. doi: 10.1161/CIRCHEARTFAILURE.111.000077. Epub 2013 Mar 21. PMID 23519586